CLINICAL TRIAL: NCT05265208
Title: A Multicenter Open-label Randomized Controlled Prospective Phase II Study Evaluating the Efficacy of Selective Internal Radiation Therapy (Yttrium-90 Glass Microspheres) Combined With Capecitabine in the Neoadjuvant Setting of Operable Intrahepatic CHOlangiocarcinoma
Brief Title: Selective Internal Radiation Therapy and Capecitabine (Chemotherapy) Treatment for Liver Cancer
Acronym: SIROCHO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-32-005; 2021-001575-16 (EudraCT Number)
Record Dates: First submitted 2022-01-25; First posted 2022-03-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Resectable Intrahepatic Cholangiocarcinoma
Keywords: Selective Internal Radiation Therapy
MeSH Terms: interventions — Capecitabine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine combined with SIRT (Experimental): Patients in the experimental arm will be treated with capecitabine combined with Selective Internal Radiotherapy (SIRT) before surgery.
  Interventions: Drug: Capecitabine; Device: Selective Internal Radiotherapy (SIRT); Procedure: Surgery
- Surgery only (Other): Patients in the control group will receive surgery only.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will given at 1250mg/m², 2 times a day with an interval of about 12 hours between two intakes, 2 weeks on, 1 week off, for 4 pre-surgery cycles.
  Other Names: L01BC06
  Arms: Capecitabine combined with SIRT
Device: Selective Internal Radiotherapy (SIRT) — During the first week of cycle 2 of capecitabine, patients will receive SIRT using Yttrium-90 glass microspheres. Treatment with Yttrium-90 glass microspheres requires two steps, one or two weeks apart. Both stages are performed under local anesthesia after a short hospitalization : the treatment simulation and therapeutic angiography.
  Arms: Capecitabine combined with SIRT
Procedure: Surgery — Surgery will be performed according to local practice.

SUMMARY:
Treatment of intrahepatic cholangiocarcinoma (ICC) remains difficult. Many patients have unresectable tumors, and survival after resection was only slightly improved with the use of adjuvant capecitabine. One of the major prognostic factors is the resection margin, patients with invaded (R1) or narrow (<5mm) margins having a higher risk of recurrence.

Selective Internal Radiation Therapy (SIRT) with Yttrium-90 microspheres (also known as SIRT) is an interesting treatment in unresectable ICC. In a phase 2 study, the investigators showed a response rate of 39% and a disease control rate of 98%. Interestingly, 9 of the 41 patients were able to see their tumors downstages to surgery. It was also recently suggested in a retrospective study that patients resected after SIRT had a better prognosis than patients that could be operated upfront, despite less favorable initial tumor characteristics.

Given the absence of validated neoadjuvant treatment, the promising activity of SIRT and chemotherapy combination in the unresectable setting, and the prognostic significance of close surgical margins, the aim of this trial is therefore to study this combination treatment in the neoadjuvant setting of resectable ICC.

DETAILED DESCRIPTION:
The study plans to randomized eligible and consent patients in two balanced parallel groups, the one defined as the experimental arm while the second consisting in the actual standard of care is defined as the control standard arm.

The experimental arm consists in 12 weeks of capecitabine combined with SIRT as neoadjuvant treatment followed by surgery. After SIRT, patients will be assessed at 10 weeks with thoracic-abdominal and pelvic CT scan and liver MRI. If the tumour is still deemed resectable, surgery will be performed at 16 weeks.

In case of discovery of contra-indication to SIRT after inclusion (such as described in the SIRT exclusion criteria section) patients will stop chemotherapy and proceed to surgery within one month. The concerned patients are still included in the study and continue the post-surgery follow-up as expected by the protocol.

In the control arm, patients will proceed to upfront surgery.

The follow - up period begins just after the surgery in both arm, and the patients are evaluated every 3 months for 2 years, then every 6 months for 3 additional years, clinically by an oncologist and radiologically with thoracic-abdominal and pelvic CT scan.

Whether progression occurred, patients will no longer be followed according to the protocol; only vital status continues to be collected until the end of the study (i.e. the last visit of the last patient).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years-old,
2. ECOG Performance Status <2,
3. Histologically-proven ICC,
4. No previous treatment for ICC,
5. Tumour deemed resectable by a hepatobiliary surgeon, validated by a Surgical Review Board,
6. Significant risk of close margins, defined as:

   1. Resection margin predicted by the surgeon <1 cm
   2. Tumour >5 cm
   3. Multifocal lesion deemed resectable, validated by a Surgical Review Board
7. Registration with a social security scheme,
8. Patient information and signature of informed consent or legal representative.

Non-inclusion Criteria:

1. Severe fibrosis (F3) ou cirrhosis (F4),
2. Inadequate haematological, hepatic, renal and coagulation functions:

   1. Haemoglobin ≤ 8,5 g/dl
   2. Neutrophils < 1,5 Giga/L
   3. Platelets < 60 Giga/L
   4. Bilirubin > 34 µmol/L
   5. ASAT/ALAT > 5 x ULN
   6. Creatinine clearance < 30 ml/min (MDRD)
   7. TP et INR > 2,3 ULN
   8. TCA > 1,5 x ULN
3. Uracil blood level >16 ng/mL,
4. Respiratory insufficiency,
5. Comorbidity precluding surgical resection, such as severe heart disease,
6. Presence of microvacuolar steatosis > 60% or regenerative nodular hyperplasia, for patients for whom a major hepatectomy is planned,
7. Contraindication to hepatic artery catheterization (vascular abnormalities, bleeding diathesis),
8. Previous chemotherapy (including for another cancer),
9. Previous abdominal (supra-mesocolic) radiotherapy (including for another cancer),
10. Other invasive malignancies,
11. Patient participate to an interventional study that tests another medical intervention before surgery,
12. Pregnant woman or likely to be or breastfeeding, or male or female patients of reproductive potential without effective contraception from screening to 30 days after the end of the treatment adjuvant,
13. Minors, individual deprived of liberty, or under any kind of guardianship,
14. Patients unable to submit to medical follow-up of the study for social, medical or psychological reasons.

Exclusion Criteria:

1. Pulmonary shunt with dose >30Gy,
2. Digestive shunting, non-correctible by interventional radiology,
3. Absence of fixation of MAA in the tumour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2030-02-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of subjects with adequate surgical margins | through study completion, an average of 5 year
  The primary endpoint will be the frequency of subjects with adequate surgical margins, defined as the number of resections AND margin ≥ 5mm.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Edeline, MD, Principal Investigator — Centre de Lutte contre le Cancer Eugène Marquis
Locations (7):
- France (7):
  - Centre de Lutte contre le Cancer Eugène Marquis, Rennes, Brittany Region
  - Groupe SUD-Haut-Lévêque - Centre Hospitalier Universitaire de Bordeaux, Pessac, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Gustave Roussy, Villejuif
  - Hôpital Beaujon, Clichy, Île-de-France Region
  - Hôpital Henri - Mondor, Créteil, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No